CLINICAL TRIAL: NCT00970853
Title: The MOM Program Continuation - 8 Year Follow-up
Brief Title: MOM Program 8-Year Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: William Penn Foundation (Other)
Responsible Party: Principal Investigator, Jerilynn Radcliffe, PI, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-007041; WPF-228-08 (Other Grant/Funding Number: The William Penn Foundation)
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Child Development
Keywords: Evaluate developmental outcomes; Evaluate child cognitive, academic, and behavioral outcomes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Control group
  Interventions: Other: Control
- MOM Program home visiting (Experimental): Mixed professional support home visiting program.
  Interventions: Behavioral: MOM Program home visiting

INTERVENTIONS:
Behavioral: MOM Program home visiting — Mixed professional home visiting program.
  Arms: MOM Program home visiting
Other: Control — Control group will receive same assessment batteries at follow-up but did not receive the home visiting program.
  Arms: Control

SUMMARY:
Study measures will evaluate cognitive, academic, and behavioral outcomes for the children, school services received, and caregiver stress and depression. The main study outcome measures include cognitive status, school functioning, and behavior. Long-term outcomes will be studied in attempt to verify the 33 and 60 month significant differences found in school participation and behavior between the intervention and control groups.

DETAILED DESCRIPTION:
This study examines 8-year follow-up results from The MOM Program, a randomized controlled trial (RCT) of a mixed professional home visiting program to promote positive developmental outcomes among children in poverty. The earlier study found significant differences in both school participation and behavior among the intervention group at ages 33 and 60 months of age. Families from the original MOM Program RCT that provide informed consent will be eligible for the study when the children are 8 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Families from the original MOM RCT that participated in the 60 month evaluation
* Able to return to Philadelphia area for testing
* Parental/guardian informed consent and child assent

Exclusion Criteria:

* Children unable to complete testing due to sensory, physical, or other deficits, as determined by clinical review by study psychologist
* Caregivers unwilling to authorize the release of school information
* Non-English speaking

Ages: 94 Months to 98 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerilynn Radcliffe, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Radcliffe J, Schwarz D, Zhao H; MOM Program. The MOM Program: home visiting in partnership with pediatric care. Pediatrics. 2013 Nov;132 Suppl 2:S153-9. doi: 10.1542/peds.2013-1021O. PMID 24187118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers from high poverty areas with singleton healthy infants weighing at least 2500g with no genetic or developmental disorders were recruited from post-partum unit of an academic hospital. At child age 8-years mothers were contacted for an in office follow-up visit. 187 of 253 eligible mothers participated.
Period: Overall Study
Arm/Group | Control | MOM Program Home Visiting
Started | 89 | 98
Completed | 89 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | MOM Program Home Visiting | Total
Number analyzed (Participants) | 89 | 98 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 89 | 98 | 187
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.96 (.12) | 7.95 (.13) | 7.95 (.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 47 | 98
  Male | 38 | 51 | 89
Region of Enrollment [Number; unit: participants]
  United States | 89 | 98 | 187

OUTCOME MEASURES:

1. Primary Outcome: Woodcock-Johnson Cognitive Ability Test, 3rd Edition (WJR-III, Cog)
Description: The WJR-III, Cog measures intelligence and cognition in children and offers a recent standardization sample and updated item content. The WJR-III, Cog was selected because it includes verbal, nonverbal, and language scales and its recent standardization sample includes an appropriate proportion of children from ethnic minority, limited parent education, and Northeastern U.S. regional families.The mean test score is 100, with a standard deviation of 15. The test yields scores from 55 (worst score) to 145 (best score).
Time Frame: 8 years post original enrollment in study
Population: All were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 89.32 (12.32) | 87.62 (14.08)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — The original sample for this study (N=302) was sufficient for an 80% detection of differences in means of at least 1/2 standard deviation. This analysis presents the results of the follow-up of the original sample; p = 0.39, t-test, 2 sided — non-adjusted for multiple comparisons

2. Secondary Outcome: Woodcock-Johnson Academic Ability Test, 3rd Edition (WJR-III, Ach), Broad Reading
Description: The WJR-III, Ach, Broad Reading measures reading achievement in children and offers a recent standardization sample and updated item content. The WJR-III, Ach, Broad Reading was selected because it includes indices of reading and a recent standardization sample that includes an appropriate proportion of children from ethnic minority, limited parent education, and Northeastern U.S. regional families.The mean test score is 100, with a standard deviation of 15. The test yields scores from 55 (worst score) to 145 (best score).
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 90.92 (17.19) | 90.94 (16.33)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — In our original sample of 302, we had 80% power to detect significant differences of at least .5 standard deviation between groups; p = .99, t-test, 2 sided

3. Secondary Outcome: Woodcock-Johnson Academic Ability Test, 3rd Edition (WJR-III, Ach), Broad Math
Description: The WJR-III, Ach, Broad Math measures math academic achievement in children and offers a recent standardization sample and updated item content. The WJR-III, Ach, Math was selected because its recent standardization sample includes an appropriate proportion of children from ethnic minority, limited parent education, and Northeastern U.S. regional families. The mean test score is 100, with a standard deviation of 15. The test yields scores from 55 (worst score) to 145 (best score).
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 94.30 (16.37) | 90.80 (16.83)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.16, t-test, 2 sided

4. Secondary Outcome: Child Behavior Checklist (CBCL), Internalizing
Description: The CBCL is part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. The CBCL is administered in interview format and respondents are asked to rate 112 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child", based on the past two months. The raw scores from the 112 items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are then derived with a mean of 50 and a standard deviation of 10. Worst value is 80; best value is 30.
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 50.30 (8.85) | 49.16 (9.61)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .40, t-test, 2 sided

5. Secondary Outcome: Child Behavior Checklist (CBCL), Externalizing
Description: The CBCL is part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. The CBCL is administered in interview format and respondents are asked to rate 112 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child", based on the past two months. The raw scores from the 112 items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. The worst possible score is 80 and the best possible score is 30.
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 54.02 (10.76) | 53.12 (10.34)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .56, t-test, 2 sided

6. Secondary Outcome: Child Behavior Checklist (CBCL),Total Problems
Description: The CBCL is part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. The CBCL is administered in interview format and respondents are asked to rate 112 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child", based on the past two months. The raw scores from the 112 items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30.
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 53.22 (10.20) | 51.81 (10.00)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .34, t-test, 2 sided

7. Secondary Outcome: Teacher Rating Form (TRF), Internalizing
Description: The TRF is the companion to the CBCL and is completed by the child's teacher. The TRF measures a broad range of behavioral, emotional, and social functioning. The TRF asks teachers to rate problem behaviors and questions about receipt of educational services. Respondents are asked to rate 112 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child", based on the past two months. The raw scores from the 112 items are then compared with scores from age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. value is 80; best value is 30.
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 48.85 (9.63) | 49.21 (11.45)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .85, t-test, 2 sided

8. Secondary Outcome: Teacher Rating Form (TRF), Externalizing
Description: The TRF is the companion to the CBCL and is completed by the child's teacher. The TRF measures a broad range of behavioral, emotional, and social functioning. The TRF asks teachers to rate problem behaviors and questions about receipt of educational services. Respondents are asked to rate 112 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child", based on the past two months. The raw scores from the 112 items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Best score is 30; worst score is 80.
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 55.75 (9.86) | 54.78 (11.73)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .61, t-test, 2 sided

9. Secondary Outcome: Teacher Rating Form (TRF), Total Problems
Description: as for outcome 8
Time Frame: 8 years from study entry
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | MOM Program Home Visiting
Number analyzed (Participants) | 89 | 98
units on a scale | 53.80 (10.17) | 52.94 (12.69)
Statistical Analysis 1: Comparison: Control vs MOM Program Home Visiting; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .67, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Control | MOM Program Home Visiting
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/98
Other Adverse Events (participants affected / at risk) | 0/89 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No